CLINICAL TRIAL: NCT06249906
Title: Clinical Study of Bioceramic Materials in Bone Defect Repair
Brief Title: Efficacy of Bioceramic Materials for Bone Defects Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20231109-04
Record Dates: First submitted 2023-12-15; First posted 2024-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Bone Lesion; Cartilage Degeneration; Osteo Arthritis Knee; Bone Fracture; Bone Injury; Bone Loss
MeSH Terms: conditions — Fractures, Bone; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Commercial bone implant product Group (Active Comparator): Bone repair products in the market such as artificial bones and allogeneic bones.
  Interventions: Device: Commercial bone implant product Group
- Mirco-structured Bioceramic Group (Experimental): β-Tricalcium phosphate (β-TCP) is a material with excellent biocompatibility and osteoinduction and bone guidance properties, which can provide mechanical strength equal to or better than that of human cancellous bone.
  Interventions: Device: Mirco-structured Bioceramic Group

INTERVENTIONS:
Device: Commercial bone implant product Group — Commercial bone implant product Group with a smooth surface （without particular microstructures）.
  Arms: Commercial bone implant product Group
Device: Mirco-structured Bioceramic Group — β-tri-Calcium phosphate with microstructures such as grooves, patterns and so on.
  Arms: Mirco-structured Bioceramic Group

SUMMARY:
The purpose of this study is to demonstrate the effect of bioceramic implants on the repair of human bone defects, and to explore the application of bioceramic materials in bone defects, bone implantation, and bone fusion. The surface microstructure of β-tricalcium phosphate bioceramic implants can be effectively controlled to guide the regeneration of bones, promote the restoration of bones, accelerate the speed of recovery, and improve bone quality, which is of great clinical and social significance.

DETAILED DESCRIPTION:
The surface microstructure of β-tricalcium phosphate bioceramic implants can be effectively controlled to guide the regeneration of bones, promote the restoration of bones, accelerate the speed of recovery, and improve bone quality, which is of great clinical and social significance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily take the test and sign the informed consent form;
2. Patients aged 18-65 years old with no history of allergies;
3. Patients able to communicate well with the investigator and follow the requirements of the entire trial.

Exclusion Criteria:

1. Patients who refuse to sign the informed consent form to participate in the trial;
2. Patients who are not in the age range of 18 to 65 years;
3. Patients with diseases unsuitbale for the trial: history of allergies, severe cardiopulmonary disease, coagulation dysfunction, Alzheimer's disease, cerebral atrophy, acute phase or sequelae of cerebrovascular disease, cognitive impairment;
4. Patients in the acute phase of local or systemic bacterial infections;
5. Patients who cannot cooperate with the operation and evaluate the effect;
6. Other conditions that are considered inappropriate by the investigator to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (SF-36) | 12 months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used.
Level of bone healing | 12 months
  X-ray, CT and MRI images would be used to evaluate the efficacy of bone healing.

OTHER OUTCOMES:
Pain self-efficacy (PSEQ) | through study completion, about 12 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire, developed in the 1980s by Michael Nicholas to assess the confidence people with ongoing pain have in performing activities while in pain. The PSEQ is applicable to all persisting pain presentations.
Incidence of nonunion | through study completion, about 12 months
  A nonunion is an arrest in the fracture repair process.
Incidence of infections | through study completion, about 12 months
  If any infections happen, the experiment would be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqiang Yao, phD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No